CLINICAL TRIAL: NCT01985048
Title: Cardiometabolic Risk in the Setting of Cardiac Rehabilitation
Brief Title: Cardiometabolic Risk in Cardiac Rehab
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Health Diagnostic Laboratory, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: R2013-3102
Record Dates: First submitted 2013-11-05; First posted 2013-11-15 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood and Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Primary Objectives:

   * To characterize cardiometabolic risk factor profiles of patients entering cardiac rehab using traditional approaches (eg LDL-C) as well as a more comprehensive panel of cardiovascular and metabolic biomarkers. It is hypothesized that the comprehensive panel will identify further increased risk that would not have been detected using only traditional approaches. Specifically, it is hypothesized that a greater percentage of the cohort will be identified with "high risk" levels of LDL-P (>1100 nmol/L) and/or apoB (>80 mg/dL) than of LDL-C (>100 mg/dL). It is further hypothesized that the prevalence of elevated Lp(a) and elevated levels of inflammatory and insulin resistance markers will be higher in this cohort when compared to population norms (HDL, inc reference data).
   * To assess improvements in laboratory and lifestyle risk factors and rate of goal attainment at completion of rehab (eg 3 months). This objective is primarily descriptive, and improvements in traditional risk factors (eg LDL-C) will be compared to existing published data. Improvements in non-traditional risk factors (eg LDL-P, insulin resistance markers) in a cardiac rehab population have not been extensively investigated.
   * To determine which attributes at baseline best predicted recurrent events and re-hospitalizations assessed one year later.
2. Secondary/Developmental Objective:

   * To inform and guide development of a subsequent study protocol designed to compare outcomes associated with biomarker-guided personalized treatment plans vs. standard of care in the cardiac rehab setting.

DETAILED DESCRIPTION:
This pilot study will characterize risk factors of patients as they enter cardiac rehab, track how comprehensive biomarker profiles change during the normal course of rehab, and associate biomarkers at baseline with MACE outcomes assessed one year later. Blood draws, vitals, and patient medical histories will be collected as subjects enter rehab and at the end of the rehab program. Major adverse cardiac events will be assessed via phone interview at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Known CAD/ IHD
* Eligibility for cardiac rehab following an acute coronary event; either:

  * ST elevation myocardial infarction
  * Non ST elevation myocardial infarction
  * Angina
  * CABG

Exclusion Criteria:

* Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Representative of the ethnic population of the areas served by the respective study sites.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Cardiometabolic biomarker risk factor | Change from Baseline at 3 months

SECONDARY OUTCOMES:
Major adverse cardiovascular events | one year

CONTACTS AND LOCATIONS:
Overall Officials: Roddy P Canosa, DO, FACC, Principal Investigator; Tina Davis, CRNP, Principal Investigator; James C. Lightfoot, M.D., Principal Investigator
Locations (3):
- United States (3):
  - Holy Spirit Hospital and Health Center, Camp Hill, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Lancaster Heart & Vascular Institution, Cardiac Rehab, Lancaster, Pennsylvania

REFERENCES:
- [Background] Suaya JA, Stason WB, Ades PA, Normand SL, Shepard DS. Cardiac rehabilitation and survival in older coronary patients. J Am Coll Cardiol. 2009 Jun 30;54(1):25-33. doi: 10.1016/j.jacc.2009.01.078. PMID 19555836
- [Background] Goel K, Lennon RJ, Tilbury RT, Squires RW, Thomas RJ. Impact of cardiac rehabilitation on mortality and cardiovascular events after percutaneous coronary intervention in the community. Circulation. 2011 May 31;123(21):2344-52. doi: 10.1161/CIRCULATIONAHA.110.983536. Epub 2011 May 16. PMID 21576654
- [Background] Hammill BG, Curtis LH, Schulman KA, Whellan DJ. Relationship between cardiac rehabilitation and long-term risks of death and myocardial infarction among elderly Medicare beneficiaries. Circulation. 2010 Jan 5;121(1):63-70. doi: 10.1161/CIRCULATIONAHA.109.876383. Epub 2009 Dec 21. PMID 20026778
- [Background] Ghashghaei FE, Sadeghi M, Mostafavi S, Heidari H, Sarrafzadegan N. The effect of the cardiac rehabilitation program on obese and non-obese females with coronary heart disease. Adv Biomed Res. 2012;1:17. doi: 10.4103/2277-9175.96077. Epub 2012 May 11. PMID 23210076
- [Background] Kubilius R, Jasiukeviciene L, Grizas V, Kubiliene L, Jakubseviciene E, Vasiliauskas D. The impact of complex cardiac rehabilitation on manifestation of risk factors in patients with coronary heart disease. Medicina (Kaunas). 2012;48(3):166-73. PMID 22588350
- [Background] Martin SS, Gosch K, Kulkarni KR, Spertus JA, Mathews R, Ho PM, Maddox TM, Newby LK, Alexander KP, Wang TY. Modifiable factors associated with failure to attain low-density lipoprotein cholesterol goal at 6 months after acute myocardial infarction. Am Heart J. 2013 Jan;165(1):26-33.e3. doi: 10.1016/j.ahj.2012.10.005. Epub 2012 Nov 17. PMID 23237130
- [Background] Gitt A, Jannowitz C, Karoff M, Karmann B, Horack M, Voller H. Treatment patterns and risk factor control in patients with and without metabolic syndrome in cardiac rehabilitation. Vasc Health Risk Manag. 2012;8:265-74. doi: 10.2147/VHRM.S28949. Epub 2012 Apr 24. PMID 22566748